CLINICAL TRIAL: NCT04683874
Title: Transfer Accuracy of 3D-printed Trays for Indirect Bonding of Orthodontic Brackets
Brief Title: Transfer Accuracy of 3D-printed Indirect Bonding Trays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thorsten Gruenheid (Other)
Responsible Party: Sponsor-Investigator, Thorsten Gruenheid, Associate Professor, University of Minnesota
Organization: University of Minnesota (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 00009952
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Dental Bonding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 3D printed tray (Experimental): 3D printed tray
  Interventions: Device: 3D printed tray

INTERVENTIONS:
Device: 3D printed tray — 3D printed tray

SUMMARY:
This study evaluates the transfer accuracy of 3D-printed trays for indirect bonding of orthodontic brackets in vivo. Accurate placement of orthodontic brackets at the beginning of treatment improves treatment efficiency and shortens treatment time. Indirect bonding is a method of placing orthodontic brackets on a plaster or digital model of the dentition, followed by the transfer of these brackets to the patients' teeth using a transfer tray. Various indirect bonding methods have been developed with the aim of improved bracket positioning and reduced chair time. The success of these methods ultimately depends on how reliably the precise positioning of the brackets on the model can be transferred to the patient's teeth.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children (ages 12 years and older) who are in the permanent dentition.

Exclusion Criteria:

* Less than 12 years of age, primary or mixed dentition, or bonded orthodontic appliances present, prosthetic restorations on the facial surfaces of teeth, craniofacial anomalies, and dental anomalies such as malformation, microdontia, or severe attrition

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Transfer accuracy | At time of bonding, i.e. day 1
  Transfer accuracy expressed as difference in bracket position between setup and clinical situation, as a result of the indirect bonding procedure. These differences will include both the magnitude and the direction, and will be reported in 6 dimensions; i.e. as mesial-distal, buccal-lingual, and occlusal-gingival linear differences as well as torque, tip, and rotation angular differences. Linear differences will be expressed in millimeters, angular differences will be expressed in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No